CLINICAL TRIAL: NCT06177600
Title: TransHealthGUIDE: Transforming Health for Gender-Diverse Young Adults Using Interventions to Drive Equity
Brief Title: TransHealthGUIDE: Transforming Health for Gender-Diverse Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rena Xu, Assistant Professor of Surgery, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00046532
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Transgender Persons; Health Services for Transgender Persons; Gender Identity
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to an Immediate Arm (access to a digital platform, plus usual care) or a Deferred Arm (usual care; access to the digital platform at 6 mo). Usual care consists of access to published resources and community support organizations, if available. The list of resources will include contact information for a suicide prevention hotline. For each Arm, the intervention period will last 6 months, followed by 6 months of observation, during which access to the intervention is maintained. Assessments will be performed at baseline, 3, 6, and 12 months to document changes in mental health outcomes, and the two groups will be compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferred Access (Other): Deferred access participants will be given usual care and gain access to the digital app at 6 months. Usual care consists of access to published resources and community support organizations, if available. The list of resources will include contact information for a suicide prevention hotline.
  Interventions: Behavioral: Interactive educational digital platform for transgender and gender-diverse (TGD) young adults and caregivers
- Immediate Access (Experimental): Immediate access participants will have access to a digital app, plus usual care, after enrollment and the deployment of the app. Usual care consists of access to published resources and community support organizations, if available. The list of resources will include contact information for a suicide prevention hotline.
  Interventions: Behavioral: Interactive educational digital platform for transgender and gender-diverse (TGD) young adults and caregivers

INTERVENTIONS:
Behavioral: Interactive educational digital platform for transgender and gender-diverse (TGD) young adults and caregivers — Investigators will develop a free mobile- and web-enabled platform for TGD young adults and their caregivers that combines educational modules with high-quality, evidence-based information and interactive features. At the time of account creation, users will complete an intake survey that will be used to personalize platform features. Young adults will be asked about their goals; mental health; access to health care; degree of caregiver support; and sociodemographic characteristics. Caregivers will be asked about their goals and self-assessed level of supportiveness of their young adults.
  Users will be assigned educational modules that build knowledge and skills related to improving mental health and navigating relationships and communication with others. Both exposure to and completion of modules will be tracked.
  Other Names: THE GUIDE

SUMMARY:
This is a randomized controlled trial to test the effectiveness of an interactive educational app-based digital intervention that provides knowledge and support to transgender and gender-diverse (TGD) young adults ages 18-29 years and their caregivers. The goal of the study is to examine the effects of exposure to the app on TGD young adult mental health outcomes.

Participants will be randomized to an Immediate Arm (access to a digital platform, plus usual care) or a Deferred Arm (usual care; access to the digital platform at 6 mo). Usual care consists of access to published resources and community support organizations, if available. The list of resources will include contact information for a suicide prevention hotline. For each Arm, the intervention period will last 6 months, followed by 6 months of observation, during which access to the intervention is maintained. Assessments will be performed at baseline, 3, 6, and 12 months to document changes in mental health outcomes, and the two groups will be compared.

The investigators plan to enroll 500 TGD young adults and their caregivers, with at least 50% (250 participants) to identify as Black, Indigenous, People of Color (BIPOC) and 50% (125 TGD young adults, 125 caregivers) to be young adult-caregiver dyads.

Ongoing process reassessments will be performed to maximize effectiveness of the intervention, including focus groups and in-depth interviews with TGD young adults, caregivers, and providers, as well as analysis of data collected through the digital platform and participant surveys. Investigators will account for sociodemographic characteristics such as race and ethnicity, age, gender identity, education status, existing mental health conditions, and history of suicidal ideation or attempt. Data will be analyzed across racial minority groups to ensure that the intervention is effective for all racial minorities; if there are discrepancies in effectiveness, additional mixed methods evaluation will be performed to identify and address potential causes.

DETAILED DESCRIPTION:
The investigators anticipate at least 80% retention across 12 mo of follow-up. This will allow detection of a reduction in suicidal ideation (primary outcome) from 40% at baseline to 26.3% or lower at 12-mo follow-up, as well as changes in the rate of psychological distress and anxiety (secondary outcome). Changes in perceptions of caregiver support and communication will also be assessed, as these are key mechanisms by which the study proposes to improve mental health outcomes. Data analysis will be performed according to intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Gender diverse individuals aged 18-29 years residing in California, Oregon, Illinois, Maryland, District of Columbia, Vermont, Connecticut, Massachusetts, Michigan, New Jersey, or New York
* Caregivers of gender diverse individuals aged 18-29 years residing in California, Oregon, Illinois, Maryland, District of Columbia, Vermont, Connecticut, Massachusetts, Michigan, New Jersey, or New York

Exclusion Criteria:

* Inability to speak, read, and write English
* Lack of device with Internet access
* Current residence in location other than California, Oregon, Illinois, Maryland, District of Columbia, Vermont, Connecticut, Massachusetts, Michigan, New Jersey, or New York

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Young adult participants between the ages of 18-29 must identify as transgender or gender expansive.
Enrollment: 500 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline, 3, 6, and 12 months
  Measure of past 3-month suicidality. Presence or absence of past 3-month suicidal ideation and risk.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 3, 6, and 12 months
  Measure of past 2-week depression. Score range is 0-27 (higher scores indicate greater degree of depressive symptoms in past 2 weeks). Score >=10 clinically elevated depressive symptoms.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 2-item (GAD-2) | Baseline, 3, 6, and 12 months
  Measure of past 2-week anxiety. Score range is 0-6 (higher scores indicate higher degree of anxious symptoms in past 2 weeks). Score >=3 clinically elevated anxiety symptoms.
SOARS Model of Non-suicidal Self-Injury | Baseline, 3, 6, and 12 months
  Measure of non-suicidal self-injury. Presence or absence of past 3-month non-suicidal self-injury.
TransFATE Family Acceptance Scale | Baseline, 3, 6, and 12 months
  Measure of family acceptance. Score range is 0-36 (higher scores indicate higher degree of family acceptance).
Family Adaptability and Cohesion Scale (FACES IV), Family Communication Subscale | Baseline, 3, 6, and 12 months
  Measure of family communication. Score range is 0-32 (higher scores indicate higher degree of family communication).
Family Adaptability and Cohesion Scale (FACES IV), Family Satisfaction Subscale | Baseline, 3, 6, and 12 months
  Measure of family satisfaction. Score range is 0-32 (higher scores indicate higher degree of family satisfaction).
Child-Parent Relationship Scale (CPRS) | Baseline, 3, 6, and 12 months
  Measure of family relationship closeness. Score range is 0-24 (higher scores indicate higher degree of closeness).
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, 3, 6, and 12 months
  Measure of social support. Score range is 0-36 (higher scores indicate more support).

CONTACTS AND LOCATIONS:
Overall Officials: Rena Xu, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reisner SL, Cole SW, Keuroghlian AS, Katz-Wise SL, Morrow C, Kane K, Feng C, Xu R. Transforming Mental Health for Transgender and Gender-Diverse Young Adults Using Interventions to Drive Equity (TransHealthGUIDE): Protocol for a Digital Randomized Controlled Trial. JMIR Res Protoc. 2025 Nov 11;14:e78619. doi: 10.2196/78619. PMID 41218206